CLINICAL TRIAL: NCT04121689
Title: Time-dependent Regulation of Postprandial Muscle Protein Synthesis After Milk Protein Ingestion in Young Men
Brief Title: Time Course of Postprandial Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14234
Record Dates: First submitted 2019-09-03; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-08

CONDITIONS: Muscle Protein Synthesis; Protein Metabolism
Keywords: Protein; Amino Acids; Anabolic Signaling; Muscle Mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Milk Protein Concentrate (Experimental): Seven young men (age: 22±1 y) will undergo repeated blood and biopsy sampling during primed continuous L-[ring-2H5]phenylalanine and L-[1-13C]leucine tracer infusions, and ingested 38 g of L-[1-13C]phenylalanine- and L-[1-13C]leucine-labeled milk protein concentrate
  Interventions: Dietary Supplement: Milk Protein Concentrate

INTERVENTIONS:
Dietary Supplement: Milk Protein Concentrate — The macronutrient composition and energy of the milk protein beverage provided to participants is 38 g protein (3.46 g leucine), 4.17 g carbohydrate, and 1.4 g fat. The milk protein met all chemical and bacteriologic specifications for human consumption. The L-[1-13C]phenylalanine and L-[1-13C]leucine enrichments in the milk protein concentrate averaged 38.3 and 10.8 mole percent excess (MPE), respectively.

SUMMARY:
The anabolic action of 'fast' whey protein on the regulation of postprandial muscle protein synthesis has been established to be short-lived in healthy young adults. Our aim was assess the time course of anabolic signaling events and stimulation of muscle protein synthesis rates (MPS) after ingestion of a food source that represents a more typical meal-induced pattern of aminoacidemia, namely milk protein concentrate, in healthy young males.

ELIGIBILITY:
Inclusion criteria

* Males
* Aged between 18-35 years
* Healthy, recreationally active
* BMI < 30 kg/m2

Exclusion criteria

* Smoking
* Allergies to milk proteins
* Vegetarians
* Diagnosed GI tract diseases
* Female
* Arthritic conditions
* A history of neuromuscular problems
* Previous participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Fractional synthesis rates of myofibrillar protein | 8 hours
  Myofibrillar protein synthesis rates will be assessed during the postabsorptive period for 3 hours, and every 1-2 hours during the 5 hours after protein ingestion. This will allow us assess the timecourse of muscle protein synthesis after eating.

SECONDARY OUTCOMES:
Phosphorylation of muscle anabolic signaling | 8 hours
  Phosphorylation of anabolic signaling pathways (mTORC1, AKT, and P70S6K) involved in the stimulation of myofibrillar protein synthesis rates will be assessed during the postabsorptive period for 3 hours, and every 1-2 hours during the 5 hours after protein ingestion.
Exogenous rate of phenylalanine appearance | 5 hours
  Dietary derived phenylalanine availability will be measured during the 5 h postprandial phase to determine its relationship with the fractional synthesis rates of myofibrillar protein and phosphorylation of muscle anabolic signaling

CONTACTS AND LOCATIONS:
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No